CLINICAL TRIAL: NCT03963843
Title: Internet-delivered Cognitive Behavioural Therapy for Persons With Spinal Cord Injury: Randomized Controlled Trial
Brief Title: Internet-delivered Cognitive Behavioural Therapy for Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-020
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries; Anxiety; Depression
Keywords: spinal cord injuries; anxiety; depression; internet-delivered cognitive behaviour therapy
MeSH Terms: conditions — Spinal Cord Injuries; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCI internet delivered cognitive behavioural therapy (Experimental): An 8-week internet- delivered cognitive behavioural therapy (ICBT) will be delivered to participants who have sustained a spinal cord injury. In addition to the online program, a health educator with experience delivering ICBT will provide support by email once a week. The health educator will spend approximately 15 minutes per week/per client.
  Interventions: Behavioral: Guided ICBT
- SCI rehabilitation mental health education (Active Comparator): Participants will receive information provided to SCI patients in usual care at specialized SCI rehabilitation units (the Spinal Cord Injury Rehabilitation Evidence (SCIRE) Community handouts available at: https://scireproject.com/community/handouts/). The lessons will include information on spinal cord injury rehabilitation: 1)spinal cord injury basics, 2)mental health after SCI, 3)pain after SCI, 4)understanding rehabilitation 5)summary of lessons through an online platform over 8 weeks. A health educator will check in with participants once a week to answer any content related questions. The health educator will spend approximately 15 minutes per week/per client.
  Interventions: Other: SCI rehabilitation mental health education

INTERVENTIONS:
Behavioral: Guided ICBT — An 8-week internet- delivered cognitive behavioural therapy (ICBT) will be delivered to participants who have sustained a spinal cord injury. In addition to the online program, a health educator with experience delivering ICBT will provide support by email once a week. The health educator will spend approximately 15 minutes per week/per client.
  Arms: SCI internet delivered cognitive behavioural therapy
Other: SCI rehabilitation mental health education — Participants will receive information provided to SCI patients in usual care at specialized SCI rehabilitation units (the Spinal Cord Injury Rehabilitation Evidence (SCIRE) Community handouts available at: https://scireproject.com/community/handouts/). The lessons will include information on spinal cord injury rehabilitation: 1)spinal cord injury basics, 2)mental health after SCI, 3)pain after SCI, 4)understanding rehabilitation 5)summary of lessons through an online platform over 8 weeks. A health educator will check in with participants once a week to answer any content related questions. The health educator will spend approximately 15 minutes per week/per client.
  Arms: SCI rehabilitation mental health education

SUMMARY:
In Canada the prevalence of spinal cord injury (SCI) is approximately 85,556, with incidence rates of traumatic and non-traumatic SCI at 1,785 and 2,286 cases per year, respectively. Common secondary health conditions experienced by individuals with SCI include psychological distress and pain. Appropriate management of these secondary conditions, through a multidisciplinary approach, is imperative as they have been shown to contribute to slower recovery, increased negative outcomes, and greater rates of rehospitalizations and health care utilization. However, resource limitations can restrict the ability of service providers to deliver these integrative biopsychosocial approaches in the community. Guided internet delivered cognitive behavioural therapy (ICBT) program offers an alternative approach for psychosocial service delivery in the community. The program provides online structured self-help modules based on the principles of cognitive behavioural therapy (CBT) in combination with guidance from a coach through weekly emails and telephone calls. ICBT was shown to have similar effects to face-to-face CBT. Results from the investigator's pilot pre-post study (ClinicalTrials.gov: NCT03457714), found significant effects of guided ICBT on primary outcome of depression (d=1.20, p=.02) post-intervention and gains were maintained at 3-month follow-up among persons with SCI. Significant improvements in secondary outcomes including pain interference, resilience, positive affect, self-efficacy, ability to participate, and grief were also found.These studies demonstrate that guided ICBT is a safe and effective alternative to face-to-face interventions and it may be beneficial for underserviced populations.

In the proposed trial, the investigators will examine the efficacy of the Guided ICBT Chronic Conditions Course for persons with SCI versus an online SCI Rehabilitation Education program. All participants will complete questionnaires prior to the start of the program, before each lesson of the program, once they have completed the program, and 3 months after completing the program. The primary outcome measures include anxiety and depression. As part of the battery of questionnaires administered after the completion of the program, clients will be asked to rate the program content, the overall service, and their satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* residing in Canada
* endorsing symptoms of anxiety or depression
* diagnosed with a spinal cord injury
* condition does not impact ability to complete treatment (ex.cognitive impairment)
* able to access a computer and internet service
* willing to provide a physician as emergency contact

Exclusion Criteria:

* high suicide risk
* suicide attempt or hospitalization in the last year
* primary problems with psychosis, alcohol or drug problems, mania
* currently receiving active psychological treatment for anxiety or depression
* not present in country during treatment
* concerns about online therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in depression | baseline, 8 weeks, 3 months, 6 months
  Measured by Patient Health Questionnaire - 9 Item (PHQ-9), Higher scores indicate greater levels of depression. 0-4 No Depression, 5-9 Mild, 10-14 Moderate, 15-19 Moderately Severe, >19 Severe
Change in anxiety | baseline, 8 weeks, 3 months, 6 months
  Measured by Generalize Anxiety Disorder - 7 Item (GAD7), higher scores indicate greater level of anxiety. 0-4 Minimal, 5-9 Mild, 10-14 Moderate, 15-21 Severe

SECONDARY OUTCOMES:
Change in psychological distress | baseline, 8 weeks, 3 months, 6 months
  Measured by Kessler 10-Item Scale, higher scores indicate greater level of distress, scores range 10-50
Change in disability | baseline, 8 weeks, 3 months, 6 months
  Measured by World Health Organization Disability Assessment Schedule - 12 Item, higher scores indicate greater level of disability. Scores range from 0-48.
Change in quality of life symptoms: SCI-QoL-SF | baseline, 8 weeks, 3 months, 6 months
  Spinal Cord Injury Quality of Life Short Form; SCI-QoL-SF, subscales of positive affect, resilience, self esteem higher scores indicate better function; subscale of grief/loss higher scores indicate severe symptoms.
Change in pain: Brief Pain Inventory-Short Form | baseline, 8 weeks, 3 months, 6 months
  Measured by Brief Pain Inventory-Short Form, the measure includes 4 items regarding pain intensity with scores ranging from 0-10 with higher scores indicating greater level of pain intensity; 7 items assess pain interference, scores ranging from 0-10 with higher scores indicating greater pain interference.
Treatment credibility | baseline and 8 weeks
  Measured by Treatment Credibility Questionnaire (TCQ) which contains 4 items. The first three items range from 0-9 with higher scores indicating better outcome, and the fourth item ranges from 0-100%, with higher scores indicating greater improvement in functioning.
Treatment satisfaction: Internet-CBT Treatment Satisfaction Measure | baseline and 8 weeks
  Measured by Internet-CBT Treatment Satisfaction Measure, each item is measured on a 0-4 scale, with higher scores indicating greater level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina; Swati Mehta, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (2):
- Canada (2):
  - Lawson Health Research Institute, London, Ontario
  - Online Therapy Unit, University of Regina, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No